CLINICAL TRIAL: NCT03121222
Title: N-acetylcysteine Supplementation in Individuals With Low Glutathione Levels: the Effects on Physical Performance and Redox Homeostasis
Brief Title: The Effects of N-acetylcysteine on Performance and Redox Homeostasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: National and Kapodistrian University of Athens (Other); European University Cyprus (Other)
Responsible Party: Principal Investigator, Vassilis Paschalis, Assistant Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 83022/2015
Record Dates: First submitted 2017-04-06; First posted 2017-04-20 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Glutathione Metabolism Anemias
MeSH Terms: interventions — Acetylcysteine; Lactose

STUDY DESIGN:
Who Masked: Participant
Masking Description: Double blind crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactose (Placebo Comparator): The placebo group received orally two lactose tablets per day for 30 days. Each individual received the capsules pre-packed in daily doses labeled with the day of consumption.
  Interventions: Drug: Lactose
- N-acetylcysteine (Experimental): The antioxidant group received orally two N-acetylcysteine tablets (each tablet contained 600 mg of NAC; Lamberts Health Care Ltd, Kent, United Kingdom). The participants were instructed to receive the capsules every twelve hours in order to achieve high concentration of N-acetylcysteine throughout the 24 h. Each individual received the capsules pre-packed in daily doses labeled with the day of consumption.
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — The antioxidant group received orally two N-acetylcysteine tablets (each tablet contained 600 mg of NAC; Lamberts Health Care Ltd, Kent, United Kingdom). The participants were instructed to receive the capsules every twelve hours in order to achieve high concentration of N-acetylcysteine throughout the 24 h. Each individual received the capsules pre-packed in daily doses labeled with the day of consumption. The supplementation period was 30-day for N-acetylcysteine.
  Arms: N-acetylcysteine
Drug: Lactose — The placebo group received orally two lactose tablets per day. The participants were instructed to receive the capsules every twelve hours. Each individual received the capsules pre-packed in daily doses labeled with the day of consumption. The supplementation period was 30-day for placebo.
  Arms: Lactose

SUMMARY:
The main objective of the present study was to investigate whether N-acetylcysteine supplementation in individuals with low glutathione levels would confer ergogenic effects by replenishing glutathione levels and by reducing oxidative stress. Towards this aim, investigators sought to exploit the large inter-individual variability in redox biomarker levels. More specifically, investigators screened 100 male participants for glutathione baseline levels in blood and formed three stratified groups according to this value (i.e., low, moderate and high; 12 individuals per group). After by-passing the regression to the mean artefact by performing a second glutathione measurement in the three aforementioned groups, investigators assessed both aerobic and anaerobic physical performance in order to acquire a more comprehensive view about the ergogenic effectiveness of the antioxidant treatment. This was accomplished by implementing three different whole-body physical performance tests (i.e., VO2max test, time trial and Wingate), as opposed to most in vivo studies that either applied isolated body-part exercise tests (e.g., by isokinetic dynamometry) or performed a single exercise test (e.g., time-to-fatigue test). It was hypothesised, that data of the present investigation will bridge the chasm between the scientific (i.e., chronic antioxidant supplementation blunts exercise performance and adaptations) and the community-based (i.e., free radicals should anyway be counteracted by "protective" exogenous antioxidants) truths about the role of antioxidants as ergogenic aids. It was also hypothesised that the results will show that low glutathione levels are linked to decreased aerobic and anaerobic physical performance accompanied by increased levels of oxidative stress and that N-acetylcysteine supplementation will restore both performance and redox homeostasis. Based on the findings of the present investigation, the widespread routine practice of consuming antioxidants during exercise training could be changed and the consumption of antioxidants would be restricted only for those who are deficient in glutathione.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects who participated recreationally in physical activities less than 3 times per week.

Exclusion Criteria:

* Subjects were excluded from the study, if they reported any musculoskeletal injury that would limit their ability to perform the exercise sessions. Participants were asked to recall whether they had participated in regular resistance or aerobic training or in unaccustomed exercise during the period before the study entry. Individuals who reported such activities were precluded from the study. Smoking and consumption of antioxidant supplements the days prior to the study were additional exclusion criteria.

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Study was limited to males in order to avoid any interference with the hormonal fluctuations during the menstrual cycle.
Enrollment: 36 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2016-02-15 (Actual); Study Completion 2016-09-12 (Actual)

PRIMARY OUTCOMES:
Measurement of maximal oxygen consumption (ml/kg/min) | 64 days
  Maximal oxygen consumption was assessed (using incremental cycling test to volitional exhaustion) on cycle ergometers (Monark, Vansbro, Sweden). Briefly, after a 5-min warm-up period at 100W, workload increased by 50W every 2.5 minutes until heart rate reached 160 bpm. Then, workload increased by 25W every 2.5 minutes until exhaustion. Respiratory gas variables were measured using a metabolic cart (Quark b2, Cosmed, Italy), which was calibrated before each test using standard gases of known concentration.
  Maximal oxygen consumption along with time trial and wingate test were used for assessing both aerobic and anaerobic physical performance in order to acquire a more comprehensive view about the ergogenic effectiveness of the antioxidant treatment.

SECONDARY OUTCOMES:
Measurement of glutathione levels (μmol/g Hb) | 64 days
  Erythrocyte GSH was determined spectrophotometrically. 20 μL of erythrocyte lysate treated with 5% TCA mixed with 660 μL of67 mMsodium potassium phosphate (pH 8.0) and 330 μL of 1mM 5,5- dithiobis-2 nitrobenzoate. The samples were incubated in the dark at room temperature for 45 min, and the absorbance was read at 412 nm.
  The measurement of glutathione was used for assessing the efficacy of NAC supplementation to restore glutathione levels in the low-glutathione group as well as the effects of NAC supplementation in the medium and high glutathione groups.

CONTACTS AND LOCATIONS:
Overall Officials: Michalis Nikolaidis, PhD, Study Director — Aristotle University Of Thessaloniki
Locations (3):
- European University Cyprus, Nicosia, Cyprus
- Greece (2):
  - National and Kapodistrian University of Athens, Athens
  - Aristotle University of Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Margaritelis NV, Theodorou AA, Paschalis V, Veskoukis AS, Dipla K, Zafeiridis A, Panayiotou G, Vrabas IS, Kyparos A, Nikolaidis MG. Experimental verification of regression to the mean in redox biology: differential responses to exercise. Free Radic Res. 2016;50(11):1237-1244. doi: 10.1080/10715762.2016.1233330. Epub 2016 Oct 25. PMID 27596985
- [Background] Jeukendrup A, Saris WH, Brouns F, Kester AD. A new validated endurance performance test. Med Sci Sports Exerc. 1996 Feb;28(2):266-70. doi: 10.1097/00005768-199602000-00017. PMID 8775164
- [Background] Paschalis V, Theodorou AA, Kyparos A, Dipla K, Zafeiridis A, Panayiotou G, Vrabas IS, Nikolaidis MG. Low vitamin C values are linked with decreased physical performance and increased oxidative stress: reversal by vitamin C supplementation. Eur J Nutr. 2016 Feb;55(1):45-53. doi: 10.1007/s00394-014-0821-x. Epub 2014 Dec 20. PMID 25526969
- [Background] Nikolaidis MG, Kyparos A, Spanou C, Paschalis V, Theodorou AA, Panayiotou G, Grivas GV, Zafeiridis A, Dipla K, Vrabas IS. Aging is not a barrier to muscle and redox adaptations: applying the repeated eccentric exercise model. Exp Gerontol. 2013 Aug;48(8):734-43. doi: 10.1016/j.exger.2013.04.009. Epub 2013 Apr 28. PMID 23628501